CLINICAL TRIAL: NCT04803708
Title: A Double-Blind and Randomized Study to Determine the Safety and Tolerability of Multiple Doses of TP-102 in Subjects With Non-Infected and Infected Diabetic Foot Ulcers
Brief Title: Bacteriophage Therapy TP-102 in Diabetic Foot Ulcers
Acronym: REVERSE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Technophage, SA (Industry)
Collaborators: VectorB2B (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TP-102_101
Record Dates: First submitted 2021-03-02; First posted 2021-03-18 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Diabetic Foot Ulcer; Pseudomonas Aeruginosa Infection; Staphylococcus Aureus Infection; Acinetobacter Infection
Keywords: Bacteriophage therapy
MeSH Terms: conditions — Diabetic Foot; Pseudomonas Infections; Staphylococcal Infections; Acinetobacter Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A- Cohort 1 (Experimental): 8 eligible subjects with non-infected DFU will be enrolled (Cohort 1) and receive IP three times weekly (TIW) every other day for up to one week. Of these 8 enrolled subjects, 6 subjects will be randomized to TP-102 and 2 to placebo. Subjects will be followed-up for 7 days.
  Interventions: Biological: TP-102
- Part B- Cohort 2 (Experimental): 18 subjects with a DFU with a grade 2 or 3 infection, as per PEDIS classification, and at least one bacterial strain susceptible to bacteriophage cocktail will be included in Cohort 2. Subjects will receive IP TIW, every other day, up to four weeks and will be randomized at a 2:1 randomization rate to either:
  * TP-102 q.d 3x weekly up to four weeks (n=12)
  * Placebo q.d. 3x weekly up to four weeks (n=6)
  Subjects will be followed-up for 7 days.
  Interventions: Biological: TP-102

INTERVENTIONS:
Biological: TP-102 — One mL of IP solution will be applied topically per cm3 of target ulcer. The titer of each bacteriophage in TP 102 is 1x10^9 plaque forming units per milliliter (PFU/mL).

SUMMARY:
This is a Phase I/IIa trial designed to evaluate topical bacteriophage therapy in patients with diabetic foot ulcers.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety of a topical bacteriophage cocktail in the treatment of non infected and infected diabetic foot ulcers with Pseudomonas aeruginosa, Staphylococcus aureus and/or Acinetobacter baumanni. Patients will also be evaluated for bacterial clearance and wound reduction.

ELIGIBILITY:
Inclusion Criteria:

Both cohorts:

* Type 1 or type 2 diabetes mellitus with glycated hemoglobin (HbA1c) ≤10, 5%
* Suitable physical and mental health as determined by the investigator based on medical history and general physical examination.
* Subjects must be medically stable based on clinical laboratory tests, medical history and vital signs. Clinical laboratory tests should be within normal values or not clinically significant, unless directly related to the condition of diabetes.
* Female subjects must fulfil one of the following criteria:

  1. At least 1 year post-menopausal (amenorrhea >12 months prior to screening);
  2. Surgically sterile (bilateral oophorectomy or hysterectomy);
  3. If of childbearing potential, must agree to use a highly effective method of birth control from screening until 14 days after the last administration of IP.
* Female subjects of childbearing potential must have a negative pregnancy test at screening.
* Male subjects with a female partner of child-bearing potential or pregnant partner must agree to use a condom from screening until 14 days after the last IP application.
* ICF signed voluntarily before any study-related procedure is performed, indicating that the subject understands the purpose of, and procedures required for the study and is willing to participate in the study.

Part A:

- Non-infected diabetic foot ulcer perfusion grade 1, depth grade 1 and infection grade 1 according to PEDIS classification.

Part B

* Infected diabetic foot ulcer meeting perfusion grade 1 or 2, depth grade 1 or 2 and infection 2 or 3,except if presence of abscess, fasciitis, osteomyelitis, and septic arthritis, according to PEDIS definition.
* Infected with at least one bacterial strain susceptible to bacteriophage cocktail assessed from culture.

Exclusion Criteria:

Both cohorts:

* Study ulcer less than 2 cm away from other ulcers in case of multiple ulcers.
* History in the 5 previous years of any cancer requiring systemic chemotherapy or radiation.
* A condition that, in the opinion of the Investigator, could compromise the well being of the subject or course of the study, or prevent the subject from meeting or performing any study requirements.
* Immunocompromised subjects due to illness, organ transplant, or immune suppressive therapies (e.g. oral or parental corticosteroids, methotrexate, immune modulators) 3 months prior to screening. Ad hoc low dose inhaled corticosteroids or topical corticosteroids are not allowed from 2 weeks prior to randomization.
* Being pregnant or breastfeeding.
* Currently participating in another clinical trial or having participated in a previous clinical trial with receipt of an investigational product within 30 days of the first administration of IP or 5 half-lives, whichever is longer.
* Subjects that, in the opinion of the Investigator or their treating physician, are dependent of the following therapies for their ulcer treatment:

  * Topical antimicrobial treatment (including isobetadine gel/dressing, silver nitrate dressing, topical antibiotic)
  * Enzymatic, autolytic, maggot debridement
  * Any active wound healing products (e.g., Dermagraft, Apligraf, Regranex, or Tegaderm hydrogel or others.)
  * Physical or cleansing modalities, antiseptics, corticosteroids, growth factors, solutions other than sterile normal saline and ulcer treatments.

Part A:

- Clinically infected ulcers

Part B:

* Suspected or confirmed abscess, fasciitis, osteomyelitis or septic arthritis.
* Subjects meeting grade 3 or above PEDIS perfusion criteria
* Planed or anticipated surgery after screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-08-07 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
1. Incidence and severity of treatment-emergent solicited local and systemic AEs and relationship to IP from first administration until 1 week after end of treatment (EOT) (end of study -EOS) | 1 week
  Local AEs include erythema/redness, swelling/induration, pain and tenderness Systemic AEs include fatigue, myalgia, fever, headache and gastrointestinal symptoms (nausea, vomiting, diarrhea)
2. Incidence and severity of treatment-emergent unsolicited AEs and relationship to IP from first administration until EOS. | 1 week
3. Incidence and severity of treatment-emergent SAEs and relationship to IP from first administration until EOS. | 1 week

SECONDARY OUTCOMES:
Proportion of subjects with significant reduction or eradication from baseline in microbiologic data via culture (cfu) at d3, d8, d15, d22, d26 and EOS | 35 days
Time (days) to significant reduction or eradication of target bacteria via culture. | 35 days
Changes in wound/ulcer healing from to baseline in terms of wound size and depth (cm^3) at EOT. | 35 days
Changes in wound/ulcer healing from to baseline in terms of wound complete closure and partial closure (25%, 50% and 75%) at EOT. | 35 days

CONTACTS AND LOCATIONS:
Overall Officials: Ran Nir-Paz, MD, Principal Investigator — Hadassah Medical Organization; Ronen Ben Ami, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (2):
- Israel (2):
  - Hadassah Medical Center, Ein Kerem, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nir-Paz R, Onallah H, Dekel M, Gellman YN, Haze A, Ben-Ami R, Braunstein R, Hazan R, Dror D, Oster Y, Cherniak M, Attal F, Barbosa AR, Dordio H, Wagner A, Jones-Dias D, Neves J, Barreto M, Leandro C, Corte-Real S, Garcia M. Randomized double-blind study on safety and tolerability of TP-102 phage cocktail in patients with infected and non-infected diabetic foot ulcers. Med. 2025 May 9;6(5):100565. doi: 10.1016/j.medj.2024.11.018. Epub 2024 Dec 30. PMID 39740667